CLINICAL TRIAL: NCT05929599
Title: Efficacy of Nasal-sprayed Probiotics Containing Bacillus Subtilis and Bacillus Clausii (LiveSpo Navax) in the Supportive Treatment of Pneumonia in Children Infected With Viral Respiratory Syncytial Virus (RSV) and Bacterial Co-infections
Brief Title: Efficacy of LiveSpo Navax in Supportive Treatment of Pneumonia in Children With RSV and Bacterial Co-infections
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Children's Hospital, Vietnam (Other)
Collaborators: Anabio R&D (Industry)
Responsible Party: Principal Investigator, Le Thi Hoa, Principal Investigator, Center for Pulmonology and Respiratory Care, Vietnam National Children's Hospital, National Children's Hospital, Vietnam
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HH1241; No.1241/BVNTW-HDDD (Other: Vietnam National Children's Hospital)
Record Dates: First submitted 2023-06-12; First posted 2023-07-03 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Acute Respiratory Tract Infections; Pneumonia; Respiratory Syncytial Virus (RSV)
Keywords: Respiratory Syncytial Virus (RSV); Acute Respiratory Tract Infections (ARTIs); Children; Oxy therapy; Nasal-spraying probiotics; Co-infection bacteria; Viral load; Cytokines; Bacillus spores
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Intervention Model Description: Blind, randomized, and controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: LiveSpo Navax and placebo 0.9% NaCl physiological saline are indistinguishable regarding taste and smell. The color and turbidity of LiveSpo Navax suspension are unrecognizable to investigators, nurses, patient's parents, and patients except for the PI, principal nurses, and analyzer, due to opaque plastic containers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Control group receives the routine treatment and uses 0.9% NaCl physiological saline:
  Routine treatment is as follows:
  * Treatment medications: antipyretic paracetamol, antibiotics following the treatment protocol for community-acquired pneumonia in children by the Ministry of Health, and antibiotics with susceptibility results, such as Amoxicillin, Augmentin, or Benzylpenicillin. In cases of severe pneumonia, the following antibiotics may be used: Benzylpenicillin + Gentamicin; Cephalosporins (Cefotaxime, Ceftriaxone) + Amikacin; Oxacillin, Bristopen, Vancomycin if Staphylococcal pneumonia is suspected.
  * Oxygen therapy: Indicated for all cases of severe pneumonia when SpO2 <92%. Use an oxygen mask or nasal cannula.
  Interventions: Drug: 0.9% NaCl physiological saline
- Navax (Experimental): Navax group receives the routine treatment and uses NaCl 0.9% plus B. subtilis and B. clausii at 5 billion CFU/5 mL (LiveSpo®️ Navax):
  Routine treatment is as follows:
  * Treatment medications: antipyretic paracetamol, antibiotics following the treatment protocol for community-acquired pneumonia in children by the Ministry of Health, and antibiotics with susceptibility results, such as Amoxicillin, Augmentin, or Benzylpenicillin. In cases of severe pneumonia, the following antibiotics may be used: Benzylpenicillin + Gentamicin; Cephalosporins (Cefotaxime, Ceftriaxone) + Amikacin; Oxacillin, Bristopen, Vancomycin if Staphylococcal pneumonia is suspected.
  * Oxygen therapy: Indicated for all cases of severe pneumonia when SpO2 <92%. Use an oxygen mask or nasal cannula.
  Interventions: Combination Product: LiveSpo Navax

INTERVENTIONS:
Drug: 0.9% NaCl physiological saline — Nasal-spraying 0.9% NaCl physiological saline is prepared by extracting 5 mL from 0.9% NaCl intravenous infusion 500 mL PP bottle (B.Braun, Germany, product declaration No. VD-32732-19), and then pouring it into the same opaque plastic spraying 10 mL-bottle that is used for LiveSpo Navax.
  Other Names: Registration number: VD-32723-19
  Arms: Control
Combination Product: LiveSpo Navax — In Vietnam, LiveSpo Navax is manufactured as a Class-A medical device product (Product declaration No.210001337/PCBA-HN) under manufacturing standards approved by Hanoi Health Department, Ministry of Health, Vietnam (Certificate No YT117-19) and ISO 13485:2016.
  Other Names: Registration number: No.210001337/PCBA-HN
  Arms: Navax

SUMMARY:
Respiratory syncytial virus (RSV) infection and bacterial co-infection are the most common causes of pneumonia. Currently, there is no vaccine available for RSV prevention, and the use of the antiviral medication ribavirin is not widely recommended for children. Therefore, the primary treatment approach follows the general protocol for pneumonia, and oxygen therapy is recommended for all cases of pneumonia with respiratory failure. However, in children, the treatment of RSV and bacterial pneumonia remains supportive to prevent bacterial co-infection and respiratory failure. Probiotics have emerged as promising and safe options for supporting the treatment of acute respiratory tract infections (ARTIs) and reducing dependence on antibiotics in recent years. In this study, investigators propose that the direct administration of probiotics through a nasal spray can offer rapid and effective symptomatic treatment for children with pneumonia who require oxygen therapy due to RSV and bacterial co-infections.

The aim of the study is to evaluate the effectiveness of nasal-spraying probiotics containing spores of two bacterial strains, Bacillus subtilis and Bacillus clausii (LiveSpo Navax), in preventing and supporting the treatment of severe pneumonia in children (who require oxygen therapy) caused by RSV infection and bacterial co-infection.

Study population: The sample size was 100, and the study was conducted at the Vietnam National Children's Hospital.

Description of Study Intervention: All 100 eligible patients were randomly divided into two groups (n = 50/each): Patients in the Control group received routine treatment and were administered 0.9% NaCl physiological saline 3 times/day, while the patients in the Navax group received LiveSpo Navax 3 times/day in addition to the same standard of care treatment. The standard treatment regimen typically lasts for 5-7 days, but its duration can be extended based on the severity of the patient's respiratory failure.

Study duration: 12 months.

DETAILED DESCRIPTION:
Pneumonia is a common disease in children and one of the leading causes of death in young children, especially those under 1 year old, infants, and malnourished children. According to the World Health Organization (WHO), an estimated 12.9 million children die each year, with 4.3 million (33.4%) of those deaths attributed to pneumonia. In Vietnam, the mortality rate from pneumonia is highest among respiratory diseases (75%), compared to the overall mortality rate of 30-35%. Statistics show that on average, a child can experience 3 to 5 episodes of acute respiratory infections per year, including 1 to 2 episodes of pneumonia. Respiratory syncytial virus (RSV) infection and bacterial co-infection are the leading causes of severe pneumonia, and the rate of co-infection can range from 26.3% to 43.6%. Commonly associated bacteria include Streptococcus pneumoniae, Haemophilus influenzae, Staphylococcus aureus, and Moraxella catarrhalis. These bacteria can invade the lower respiratory tract and cause secondary infections, taking advantage of respiratory damage caused by RSV.

Currently, there is no vaccine or specific treatment available for children with RSV infection, and oxygen therapy is generally recommended for children experiencing respiratory failure. The use of the monoclonal antibody palivizumab and the antiviral nucleotide drug ribavirin is considered too expensive or risky for children and is only recommended for high-risk patients. Bacterial co-infections often require antibiotic treatment based on suspected or known pathogens, but the use of antibiotics has significant side effects and raises concerns about the development of resistance.

In recent years, probiotics have gained popularity as promising and safe candidates for preventive and supportive therapies in respiratory infections, aiming to aid in the treatment and reduction of respiratory tract infections. Probiotics, which are live microorganisms providing health benefits when consumed in adequate quantities, have traditionally been used to promote gut health. However, their potential role in respiratory infections, specifically RSV pneumonia, has not been extensively explored. Some studies suggest that certain strains of probiotics can directly interact with viruses, capturing them, inducing secondary growth to inhibit virus entry and growth, or modulating the immune response to reduce the risk of respiratory infections. Nevertheless, the impact of oral probiotics on the respiratory tract of infants is typically delayed (usually around 3-12 months) and primarily used for prophylaxis rather than as an adjunct to ARTI treatment. Hence, there is a need for alternative delivery routes of probiotics in ARTI treatment. In our recent study, we have proven that the nasal-spraying Bacillus spore liquid-form probiotics (LiveSpo Navax containing > 5 billion B. subtilis ANA4 and B. clausii ANA39/ 5 mL ampoule) can rapidly and effectively relieve symptoms of ARTIs due to respiratory syncytial virus (RSV) infection while exhibiting strong impacts in reducing the viral load and inflammation. This finding is the first demonstration that spraying probiotics directly into the nose could be a quick and effective symptomatic treatment for ARTIs.

In this following study, we conducted the double-blind, randomized, and controlled clinical trial to further examine the efficacy of LiveSpo Navax in supporting the treatment of children with severe pneumonia who require oxygen therapy due to RSV and bacterial co-infections.

Methods: A randomized, blind, and controlled clinical trial will be conducted. The parents of the patients will be required to provide various information about their children, including their full name, sex, age, obstetric history, vaccination history, and antibiotic use history. After obtaining informed consent, 100 patients with severe pneumonia due to RSV and bacterial co-infection will be randomly assigned to two groups (n = 50/group): the control group (referred to as the "Control" group) will receive 0.9% NaCl physiological saline, and the experimental group (referred to as the "Navax" group) will receive the probiotics LiveSpo Navax. The patients will be given a coded spray in the form of a blind sample to ensure the objectivity of the study. Clinical follow-up will be conducted for 7 days or more, and nasopharyngeal samples will be collected on day 0 and day 3 to evaluate potential reductions in viral load, co-infection bacteria, modulation of overreacted cytokine release, and the presence of probiotic spores in the patient's nasal mucosa.

Real-time PCR will be used to detect microorganisms in the nasopharyngeal samples. Semi-quantitative assays will be performed to measure changes in RSV load and co-infection bacterial concentrations using the real-time PCR routine protocol, which has been standardized under ISO 15189:2012 criteria and is routinely used at the Vietnam National Children's Hospital. Detection of Bacillus strains belonging to B. subtilis and B. clausii will be conducted using real-time PCR SYBR Green assay, which is routinely performed at the Spobiotic Research Center in Hanoi, Vietnam.

ELISA assays will be used to quantify pro-inflammatory cytokine levels (e.g., IL-6, IL-8, TNF-alpha...) and Immunoglobulin A (IgA) levels. The assays will be performed using an ELISA kit according to the manufacturer's instructions.

Nasal microbiome analysis will be conducted using next-generation sequencing (NGS) of the 16S rRNA gene at Macrogen in Seoul, Korea, on the Illumina MiSeq platform with a 2 x 250 bp run configuration.

During the treatment, patients will be monitored daily for typical clinical symptoms of severe pneumonia due to RSV and bacterial co-infection, including runny nose, chest depression, dry rales, moist rales, oxymetry (SpO2) (%), pulse (beats/min), and breath (beats/min), as well as the number of days requiring oxygen therapy... until discharge. The patients' health conditions will be observed by doctors and nurses, and their information will be recorded in medical records. Throughout the study, parents will be asked to refrain from administering other probiotics, either via nasal spray or oral administration, and from using other 0.9% NaCl physiological saline sprays for nasal cleaning.

Data collection and statistical analysis will involve collecting individual medical records and systematically organizing the patient's information into a dataset. The efficacy of LiveSpo Navax will be evaluated and compared to 0.9% NaCl physiological saline based on various clinical and sub-clinical criteria obtained from the Navax and Control groups. These criteria include the number of days until symptomatic relief, the reduction levels (2^△Ct) of RSV load, and co-infection bacterial concentrations. The △Ct for target genes will be calculated as Ct (threshold cycle) at day 3 - Ct at day 0, while the Ct of the internal control will be adjusted to be equal among all samples. Additionally, the reduced levels of cytokines (e.g. IL-6, IL-8, TNF-alpha...), and IgA will be assessed. The tabular analysis will be performed using the χ2 test or Fisher's exact test for dichotomous variables with expected cell values below five. Continuous variables will be compared using the Wilcoxon test, t-test, or Mann-Whitney test when data are not normally distributed. The correlations among variables will be assessed using Spearman's correlation analysis. Statistical and graphical analyses will be performed using GraphPad Prism v8.4.3 software (GraphPad Software, CA, USA). The significance level for all analyses will be set at p < 0.05.

Expected outcomes: (i) LiveSpo Navax is expected to alleviate RSV infection symptoms about 25% more effectively, with 90% of patients in the Navax group being symptom-free at day 3-7 of intervention (depending on symptoms), compared to 65% of patients in the Control group; (ii) Patients in the Navax group are expected to experience more significant reductions (>10 fold) in RSV load compared to patients in the Control group on day 3 of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children (male/female) aged from 1 to 24 months.
* Hospitalization due to pneumonia.
* RSV is positive by rapid test.
* Bacterial co-infection (Yes or No).
* Oxygen therapy (Yes or No).
* Parents of the pediatric patient agree to participate in the study, explain and sign the research consent form.

Exclusion Criteria:

* Children with underlying medical conditions (congenital heart disease, airway malformation).
* Hospital-acquired pneumonia.
* Newborn babies.
* Have a history of drug allergy.
* Discharged before day 3.
* Lost to follow-up.
* Withdrawn from the trial.
* Continuing in the trial but missing data.
* Meeting the criteria for psychiatric disorders other than depression and/or anxiety.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-07-27 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with free respiratory symptoms | Day 0 to day 10
  Percentage (%) of RSV-infected patients with free respiratory symptoms including runny nose, chest depression, difficulty breathing, dry rales, and moist rales...
Number of days requiring oxygen therapy | Day 0 to day 10
  Number of days the patient requires oxygen therapy intervention.
Number of days using antibiotics | Day 0 to day 10
  Number of days the patient using antibiotics

SECONDARY OUTCOMES:
Patient's breath | Day 0 to day 3
  Monitoring the patient's breath (beat/min) on a daily basis during treatment
Patient's pulse | Day 0 to day 3
  Monitoring the patient's pulse (beat/min) on a daily basis during treatment
Patient's pulse oxygen (SpO2) | Day 0 to day 3
  Monitoring the patient's pulse oxygen - SpO2 (%) on a daily basis during treatment
Change RSV concentration | Day 0 and day 3
  Change concentration of respiratory syncytial virus in nasopharyngeal samples, as indicated by real-time PCR threshold cycle (Ct) value at day 3 (after treatment) compared with day 0 (before treatment)
Change co-infection bacterial concentrations | Day 0 and day 3
  Change concentration of Co-infection bacterial in nasopharyngeal samples, as indicated by real-time PCR threshold cycle (Ct) value at day 3 (after treatment) compared with day 0 (before treatment)
Change cytokines levels | Day 0 and day 3
  Change cytokines levels (pg/mL) (e.g., tumor necrosis factor-α (TNF-α), interleukin-6 (IL-6), interleukin-8 (IL-8) in nasopharyngeal samples at day 3 (after treatment) compared with day 0 (before treatment)
Change Immunoglobulin A (IgA) level | Day 0 and day 3
  Change IgA level (mg/mL) in nasopharyngeal samples at day 3 (after treatment) compared with day 0 (before treatment)
Change the nasal microbiota | Day 0 and day 3
  Alter the nasal microbiota, as indicated by changes in the diversity of nasal microbial species based on the data analysis of next-generation sequencing (NGS) on day 3 (after treatment) compared to day 0 (before treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Hoa T Le, MSc. MD, Principal Investigator — The Center for Pulmonology and Respiratory Care, Vietnam National Children's Hospital; Hanh TH Le, PhD. MD, Study Director — The Center for Pulmonology and Respiratory Care, Vietnam National Children's Hospital
Locations (1):
- The Center for Pulmonology and Respiratory Care, Vietnam National Children's Hospital, Hà Nội, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data or samples share that will be coded, with no PHI include. Approval of the request and execution of all applicable agreements (i.e., a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a study protocol, informed consent form (ICF), clinical study peport (CSR). For more information or to submit a request, please contact anabio.rd2021@gmail.com

REFERENCES:
- [Background] Bryce J, Boschi-Pinto C, Shibuya K, Black RE; WHO Child Health Epidemiology Reference Group. WHO estimates of the causes of death in children. Lancet. 2005 Mar 26-Apr 1;365(9465):1147-52. doi: 10.1016/S0140-6736(05)71877-8. PMID 15794969
- [Background] Benguigui Y. [Magnitude and control of acute respiratory infections in children]. Salud Publica Mex. 1988 May-Jun;30(3):362-9. Spanish. PMID 3187734
- [Background] Rudan I, Boschi-Pinto C, Biloglav Z, Mulholland K, Campbell H. Epidemiology and etiology of childhood pneumonia. Bull World Health Organ. 2008 May;86(5):408-16. doi: 10.2471/blt.07.048769. PMID 18545744
- [Background] Do AH, van Doorn HR, Nghiem MN, Bryant JE, Hoang TH, Do QH, Van TL, Tran TT, Wills B, Nguyen VC, Vo MH, Vo CK, Nguyen MD, Farrar J, Tran TH, de Jong MD. Viral etiologies of acute respiratory infections among hospitalized Vietnamese children in Ho Chi Minh City, 2004-2008. PLoS One. 2011 Mar 24;6(3):e18176. doi: 10.1371/journal.pone.0018176. PMID 21455313
- [Background] Bellos A, Mulholland K, O'Brien KL, Qazi SA, Gayer M, Checchi F. The burden of acute respiratory infections in crisis-affected populations: a systematic review. Confl Health. 2010 Feb 11;4:3. doi: 10.1186/1752-1505-4-3. PMID 20181220
- [Background] Gruber C, Keil T, Kulig M, Roll S, Wahn U, Wahn V; MAS-90 Study Group. History of respiratory infections in the first 12 yr among children from a birth cohort. Pediatr Allergy Immunol. 2008 Sep;19(6):505-12. doi: 10.1111/j.1399-3038.2007.00688.x. Epub 2007 Dec 21. PMID 18167154
- [Background] Lin HC, Liu YC, Hsing TY, Chen LL, Liu YC, Yen TY, Lu CY, Chang LY, Chen JM, Lee PI, Huang LM, Lai FP. RSV pneumonia with or without bacterial co-infection among healthy children. J Formos Med Assoc. 2022 Mar;121(3):687-693. doi: 10.1016/j.jfma.2021.08.012. Epub 2021 Aug 24. PMID 34446339
- [Background] Bakaletz LO. Viral-bacterial co-infections in the respiratory tract. Curr Opin Microbiol. 2017 Feb;35:30-35. doi: 10.1016/j.mib.2016.11.003. Epub 2016 Dec 7. PMID 27940028
- [Background] van den Bergh MR, Biesbroek G, Rossen JW, de Steenhuijsen Piters WA, Bosch AA, van Gils EJ, Wang X, Boonacker CW, Veenhoven RH, Bruin JP, Bogaert D, Sanders EA. Associations between pathogens in the upper respiratory tract of young children: interplay between viruses and bacteria. PLoS One. 2012;7(10):e47711. doi: 10.1371/journal.pone.0047711. Epub 2012 Oct 17. PMID 23082199
- [Background] Aston SJ. Pneumonia in the developing world: Characteristic features and approach to management. Respirology. 2017 Oct;22(7):1276-1287. doi: 10.1111/resp.13112. Epub 2017 Jul 6. PMID 28681972
- [Background] Friedman JN, Rieder MJ, Walton JM; Canadian Paediatric Society, Acute Care Committee, Drug Therapy and Hazardous Substances Committee. Bronchiolitis: Recommendations for diagnosis, monitoring and management of children one to 24 months of age. Paediatr Child Health. 2014 Nov;19(9):485-98. doi: 10.1093/pch/19.9.485. PMID 25414585
- [Background] Pochon C, Voigt S. Respiratory Virus Infections in Hematopoietic Cell Transplant Recipients. Front Microbiol. 2019 Jan 9;9:3294. doi: 10.3389/fmicb.2018.03294. eCollection 2018. PMID 30687278
- [Background] Principi N, Cozzali R, Farinelli E, Brusaferro A, Esposito S. Gut dysbiosis and irritable bowel syndrome: The potential role of probiotics. J Infect. 2018 Feb;76(2):111-120. doi: 10.1016/j.jinf.2017.12.013. Epub 2017 Dec 29. PMID 29291933
- [Background] Elshaghabee FMF, Rokana N, Gulhane RD, Sharma C, Panwar H. Bacillus As Potential Probiotics: Status, Concerns, and Future Perspectives. Front Microbiol. 2017 Aug 10;8:1490. doi: 10.3389/fmicb.2017.01490. eCollection 2017. PMID 28848511
- [Background] Tran DM, Tran TT, Phung TTB, Bui HT, Nguyen PTT, Vu TT, Ngo NTP, Nguyen MT, Nguyen AH, Nguyen ATV. Nasal-spraying Bacillus spores as an effective symptomatic treatment for children with acute respiratory syncytial virus infection. Sci Rep. 2022 Jul 20;12(1):12402. doi: 10.1038/s41598-022-16136-z. PMID 35858943
- [Background] Song M, Hong HA, Huang JM, Colenutt C, Khang DD, Nguyen TV, Park SM, Shim BS, Song HH, Cheon IS, Jang JE, Choi JA, Choi YK, Stadler K, Cutting SM. Killed Bacillus subtilis spores as a mucosal adjuvant for an H5N1 vaccine. Vaccine. 2012 May 9;30(22):3266-77. doi: 10.1016/j.vaccine.2012.03.016. Epub 2012 Mar 22. PMID 22446640
- [Background] Marseglia GL, Tosca M, Cirillo I, Licari A, Leone M, Marseglia A, Castellazzi AM, Ciprandi G. Efficacy of Bacillus clausii spores in the prevention of recurrent respiratory infections in children: a pilot study. Ther Clin Risk Manag. 2007 Mar;3(1):13-7. doi: 10.2147/tcrm.2007.3.1.13. PMID 18360611
- [Background] Lehtoranta L, Pitkaranta A, Korpela R. Probiotics in respiratory virus infections. Eur J Clin Microbiol Infect Dis. 2014 Aug;33(8):1289-302. doi: 10.1007/s10096-014-2086-y. Epub 2014 Mar 18. PMID 24638909
- [Derived] Thi Le H, Thi Bich Phung T, Thi Bui H, Thi Hong Le H, Tran DM, Nguyen NH, Phan HT, Tran VD, Vu Pham U, Van Phan N, Thu Do H, Nguyen AH, Pham TD, Thi Van Nguyen A. Nasal-spraying Bacillus spore probiotics for pneumonia in children with respiratory syncytial virus and bacterial co-infections: a randomized clinical trial. Commun Med (Lond). 2025 Aug 7;5(1):336. doi: 10.1038/s43856-025-01029-9. PMID 40770421